CLINICAL TRIAL: NCT01027793
Title: Randomized Clinical Trial Comparing Treatment of Tretinoin or Superficial Dermabrasion for Recent Stretch Marks
Brief Title: Trial Comparing Treatment of Tretinoin or Superficial Dermabrasion for Stretch Marks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-CBED08-01
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Stretch Marks; Striae; Treatment
Keywords: Stretch marks; Striae; Tretinoin; Superficial dermabrasion
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tretinoin (Active Comparator): Group 1 will receive tretinoin cream 0.05%(Vitanol A, Stiefel) that should be applied daily in areas affected by stretch marks, in both sides, for a period of 16 weeks.
  Interventions: Drug: Tretinoin cream 0.005%
- Superficial Dermabrasion (Active Comparator): Group 2 will receive 16 sessions of dermabrasion that would be held in the research center.
  Interventions: Device: Superficial Dermabrasion

INTERVENTIONS:
Drug: Tretinoin cream 0.005% — Group 1 will receive tretinoin cream 0.05%(Vitanol A, Stiefel) that should be applied daily in areas affected by stretch marks, in both sides, for a period of 16 weeks.
  Other Names: (Vitanol A, Stiefel)
  Arms: Tretinoin
Device: Superficial Dermabrasion — Group 2 will receive 16 sessions of dermabrasion that would be held in the research center
  Arms: Superficial Dermabrasion

SUMMARY:
This study aims to evaluate head-to-head the effectiveness of tretinoin 0.5% and superficial dermabrasion in subjects that have recent stretch marks.

DETAILED DESCRIPTION:
Healthy female subjects, from 11 t0 25 years old, that have thin (1-5mm) recent(less than 6 months of evolution),reddish or purple line stretch marks. The striae should be symmetrical and it could be located in the abdomen,breasts, upper arms, thighs (both inner and outer), hips, and buttocks.

Thirty subjects will be randomly divided in two groups:

Group 1 will receive tretinoin cream that should be applied daily in areas affected by stretch marks.

Group 2 will receive 16 sessions of dermabrasion that would be held in the research center.

Subjects will be evaluated by pictures, measurement of width and length of stretch marks, using Mirror System(Canfield).

Biopsy to quantify alterations of epidermis and dermis of treated area, will be held pre-treatment and 2 weeks after the conclusion of treatment. For biopsy will be used a punch of 3mm.

The results will be evaluated two weeks after the conclusion of the interventions. An independent dermatologist, blinded for intervention, will analyse pictures pre and post treatment. This subjective evaluation will be performed using Global Aesthetic Improvement Scale.

Safety and adverse events will be assessed each visit.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, aged between 11 and 25 years
* Female subjects of childbearing age that present a negative urine pregnancy test and are using an effective contraceptive method for at least 3 months prior the study
* Subjects that have thin (1-5mm) recent(less than 6 months of evolution),reddish or purple line stretch marks. The striae should be symmetrical and it could be located in the abdomen,breasts, upper arms, thighs (both inner and outer), hips, and buttocks
* Subjects agreeing to take part of the study, after being fully informed of the purpose and the nature of the investigation and after having signed the informed consent form
* Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol
* Subjects who had never received treatment for striae in the studied area

Exclusion Criteria:

* Subjects whose medical history and physical examination present clinical pathology, as marfan Syndrome, cushing, systemic autoimmune or neurological diseases
* Pregnant or women in breastfeeding, or women planning to become pregnant
* Previous treatment for striae in the local area of the study.
* Subjects that are in use of tretinoin or glycolic acid in the local area of the study.
* Presence of white striae in the local area of the study
* History of Connective Tissue Disease
* History of keloid development or skin healing problems
* Subjects that are taking medications associated with striae development, as systemic corticosteroids, indinavir, hormonal replacement therapy
* Hypersensibility to retinoic acid
* Subjects who intend to get tan in the area of the study, through exposure of sun or tanning machines during the study
* Subjects that have a variation in their weight of more than 2 kg in a period of four months prior the study
* Predisposition for chronic inflammatory process
* Subjects with chronic diseases as diabetes, cardiopathy, neoplasm, HIV and autoimmune diseases (vitiligo, lupus)

Ages: 11 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Hexsel, MD, Principal Investigator — Brazilian Center For Studies in Dermatology
Locations (1):
- Brazilian Center for Studies in Dermatology, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Tretinoin: Group 1 will receive tretinoin cream 0.05% (Vitanol A, Stiefel) that should be applied daily in areas affected by stretch marks, in both sides, for a period of 16 weeks.
  Tretinoin cream 0.005%: Group 1 will receive tretinoin cream 0.05%(Vitanol A, Stiefel) that should be applied daily in areas affected by stretch marks, in both sides, for a period of 16 weeks.
Period: Overall Study
Arm/Group | Tretinoin | Superficial Dermabrasion
Started | 17 | 15
Completed | 10 | 12
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: Per protocol assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Tretinoin | Superficial Dermabrasion | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (4.3) | 17.0 (3.2) | 16.9 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 10 | 12 | 22
Fitzpatrick skin phototype [Count of Participants; unit: Participants] — Phototype I - Pale white skin, blue/green eyes, blond/red hair; Always burns, does not tan Phototype II - Fair skin, blue eyes; Burns easily, tans poorly Phototype III - Darker white skin; Tans after initial burn Phototype IV - Light brown skin; Burns minimally, tans easily Phototype V - Brown skin; Rarely burns, tans darkly easily Phototype VI - Dark brown or black skin; Never burns, always tans darkly
  Participants
    Fitzpatrick skin phototype I | 0 | 0 | 0
    Fitzpatrick skin phototype II | 4 | 5 | 9
    Fitzpatrick skin phototype III | 5 | 6 | 11
    Fitzpatrick skin phototype IV | 1 | 1 | 2
    Fitzpatrick skin phototype V | 0 | 0 | 0
    Fitzpatrick skin phototype VI | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (4.4) | 24.8 (3.3) | 24.3 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Width of Stretch Marks
Description: Striae width was measured with Mirror Medical Imaging Software (Canfield Scientific, Inc., Parsippany, NJ)
Time Frame: Baseline and 16 weeks
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Tretinoin | Superficial Dermabrasion
Number analyzed (Participants) | 10 | 12
centimeters
  Baseline | 0.199 (0.129) | 0.146 (0.052)
  Week 16 | 0.088 (0.073) | 0.077 (0.040)

2. Primary Outcome: Length of Stretch Marks
Description: Striae length was measured with Mirror Medical Imaging Software (Canfield Scientific, Inc., Parsippany, NJ)
Time Frame: Baseline and 16 weeks
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Tretinoin | Superficial Dermabrasion
Number analyzed (Participants) | 10 | 12
centimeters
  Baseline | 1.371 (0.631) | 1.518 (0.386)
  Week 16 | 0.894 (0.457) | 1.111 (0.673)

3. Secondary Outcome: Global Aesthetic Improvement Scale
Description: 1. Very much improved: Optimal cosmetic result for the implant in this patient
  2. Much improved: Marked improvement in appearance from the initial condition but not completely optimal for this patient; touch-up would slightly improve the result 3 - Improved: Obvious improvement in appearance from the initial condition, but touch-up or retreatment is indicated 4 - No change: Appearance essentially the same as the original condition 5 - Worse: Appearance worse than the original condition
Time Frame: 16 weeks
Population: Per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin | Superficial Dermabrasion
Number analyzed (Participants) | 10 | 12
Participants
  Very much improved | 3 | 1
  Much improved | 5 | 5
  Improved | 2 | 6

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction measured with Lickert scale (Very satisfied, Satisfied, Neither satisfied nor unsatisfied, unsatisfied, very unsatisfied)
Time Frame: 16 weeks
Population: Per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Tretinoin | Superficial Dermabrasion
Number analyzed (Participants) | 10 | 12
Participants
  Very satisfied | 1 | 6
  Satisfied | 4 | 4
  Neither satisfied nor unsatisfied | 1 | 2

ADVERSE EVENTS:
Arm/Group | Tretinoin | Superficial Dermabrasion
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 7/10 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tretinoin (N=10) | Superficial Dermabrasion (N=12)
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5 — Itching on the treated area.
Erythema (Skin and subcutaneous tissue disorders) | 6 | 4 — Erythema on the treated area.
Scaling (Skin and subcutaneous tissue disorders) | 4 | 2 — Scaling on the treated area
Stinging (Skin and subcutaneous tissue disorders) | 2 | 4 — Stinging on the treated area

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes